CLINICAL TRIAL: NCT00913406
Title: Effect of Lutein in S-26 Gold on Growth and Safety
Acronym: S-26 Gold L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 9041A1-902
Record Dates: First submitted 2009-05-28; First posted 2009-06-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Effect of lutein fortification growth healthy term infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Experimental=Standard formula with lutein added to the formula
  Interventions: Other: Lutein fortification
- 2 (Active Comparator): Active Comparator=Standard formula
  Interventions: Other: Standard formula

INTERVENTIONS:
Other: Lutein fortification
  Arms: 1
Other: Standard formula
  Arms: 2

SUMMARY:
Study to determine if the addition of lutein to infant formula supports healthy growth and development in healthy full term infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 0-14 days
* Full Term birth and AGA Parent(s) signed informed consent

Exclusion Criteria:

* Unhealthy infant
* Participation in other clinical trial
* Use of prohibited medications

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Weight gain/day in grams/day | 4 months

SECONDARY OUTCOMES:
Collection of adverse experiences | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer